CLINICAL TRIAL: NCT00107380
Title: Iodine-131-Labeled Monoclonal Anti-B1 Antibody (I-131 Tositumomab) in Combination With Cyclophosphamide, Doxorubicin, Vincristine, Prednisone and Rituximab Therapy for Patients ≥ Age 60 With Advanced Stage Diffuse Large B-Cell NHL: A Phase II Study
Brief Title: S0433 Iodine I 131 Tositumomab, Rituximab, and Combination Chemotherapy in Treating Older Patients With Stage II, Stage III, or Stage IV Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000415955; S0433 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine; tositumomab I-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- R-CHOP x 8 with I-131 Tositumomab (Experimental): Cyclophosphamide 750 mg/m2 IV Day 1 Doxorubicin 50 mg/m2 IV Day 1 Vincristine 1.4 mg/m2 IV Day 1 Prednisone 100 mg PO Days 1-5 Rituximab 375 mg/m2 IV Day 1 Q 21 Days x 6 cycles
  Unlabeled Anti-B1 Antibody 450 mg IV Day 170 Dosimetric dose 35 mg IV Day 170
  Unlabeled Anti-B1 Antibody 450 mg IV Day 177 Therapeutic dose 35 mg IV Day 177
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate; Radiation: tositumomab and iodine I 131 tositumomab

INTERVENTIONS:
Biological: rituximab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate
Radiation: tositumomab and iodine I 131 tositumomab

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies, such as iodine I 131 tositumomab, can find cancer cells and carry cancer-killing substances to them without harming normal cells. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin, vincristine, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving a radiolabeled monoclonal antibody together with rituximab and combination chemotherapy may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving iodine I 131 tositumomab together with rituximab and combination chemotherapy works in treating older patients with stage II, stage III, or stage IV B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 2-year progression-free survival of older patients with previously untreated bulky stage II or stage III or IV diffuse large B-cell non-Hodgkin's lymphoma treated with iodine I 131 tositumomab in combination with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone.
* Determine the response rate (partial response, complete unconfirmed response, and complete response) in patients treated with this regimen.
* Determine the 2-year progression-free survival and response rate (partial response, complete unconfirmed response, and complete response) in B-cell lymphoma 2 (BCL-2) positive patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Rituximab and chemotherapy: Patients receive R-CHOP comprising rituximab IV over 6 hours; cyclophosphamide IV over 15-45 minutes; doxorubicin IV over 5-20 minutes; and vincristine IV over 5-15 minutes on day 1 and oral prednisone on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo a restaging evaluation. Patients without progressive disease receive CHOP chemotherapy comprising cyclophosphamide, doxorubicin, vincristine, and prednisone as outlined above. Treatment with CHOP chemotherapy repeats every 21 days for 2 courses.
* Radiolabeled monoclonal antibody therapy: Approximately 4-8 weeks after completion of chemotherapy, patients receive tositumomab IV over 1 hour followed by a dosimetric dose of iodine I 131 tositumomab IV over 20 minutes. Patients then undergo gamma scans over a 1-week period in order to determine the correct treatment dose of iodine I 131 tositumomab. No more than 2 weeks after administration of the dosimetric dose, patients receive tositumomab IV over 1 hour followed by a treatment dose of iodine I 131 tositumomab IV over 20 minutes.

After completion of study treatment, patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study within 15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of diffuse large B-cell non-Hodgkin's lymphoma, meeting 1 of the following stage criteria:

  * Bulky stage II disease
  * Stage III disease
  * Stage IV disease
* Confirmed cluster of differentiation antigen 20 (CD20) antigen-positive disease
* Bidimensionally measurable disease
* Less than 20,000/mcL circulating lymphoid cells on white blood cell (WBC) differential count
* Adequate sections AND a paraffin block OR ≥ 10 unstained sections from the original diagnostic specimen available

  * Needle aspiration or cytology are not considered adequate
* No clinical evidence of central nervous system (CNS) involvement by lymphoma
* No prior diagnosis of indolent lymphoma

  * No histologic transformation

PATIENT CHARACTERISTICS:

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* Ejection fraction ≥ 45% by multiple gated acquisition scan (MUGA) OR
* No significant abnormalities by echocardiogram

Pulmonary

* No requirement for continuous supplemental oxygen

Other

* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, stage I or II cancer in complete remission, or carcinoma in situ of the cervix
* No known HIV positivity

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior antibody therapy for lymphoma

Chemotherapy

* No prior chemotherapy for lymphoma

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for lymphoma

Surgery

* No prior solid organ transplantation

Other

* Concurrent enrollment on protocol SWOG-8947 (lymphoma serum repository) or protocol SWOG-8819 (lymphoma tissue repository) is encouraged

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2005-11; Primary Completion 2013-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W. Friedberg, MD, Study Chair — James P. Wilmot Cancer Center; Richard I. Fisher, MD, Study Director — James P. Wilmot Cancer Center
Locations (78):
- United States (78):
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Falck Cancer Center at Arnot Ogden Medical Center, Elmira, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- R-CHOP + I-131-tositumomab: Patients receive cyclophosphamide 750 mg/m^2 IV over 15 minutes, doxorubicin 50 mg/m^2 IV, and vincristine IV on days 1, 22, 43, 64, 85, 106, 127, and 148. Patients also receive oral prednisone 100 mg daily on days 1-5, 22-26, 43-47, 64-68, 85-89, 106-110, 127-131, and 148-152; rituximab 375 mg/m^2 IV on days 1, 22, 43, 64, 85, and 106; unlabeled anti-B1 antibody 450 mg/m^2 IV and dosimetric dose 35 mg IV over 20 minutes on day 170, and unlabeled anti-B1 antibody 450 mg IV and therapeutic dose 35mg IV over 20 minutes on day 177.
Period: Overall Study
Arm/Group | R-CHOP + I-131-tositumomab
Started | 86
Eligible | 84
Completed | 56
Not Completed | 30
Not completed — Adverse Event | 7
Not completed — Refusal Unrelated to Adverse Event | 7
Not completed — Progression/relapse | 4
Not completed — Death | 3
Not completed — Other - not protocol specified | 7
Not completed — Ineligible | 2

BASELINE CHARACTERISTICS:
Population: All eligible patients who started treatment were included in the analysis
Arm/Group | R-CHOP + I-131-tositumomab
Number analyzed (Participants) | 84
Age, Continuous [Median (Full Range); unit: years] | 63.8 [29.9 to 85.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 65
  Unknown or Not Reported | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 78
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) at 2 Years
Description: Clinical responses were evaluated according to International Workshop NHL criteria (Cheson et al, 1999). Progression disease was defined as if a (CR, CRU) was not achieved at a previous assessment, a 50% increase in the SPD of target measurable lesions over the smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline. Appearance of a new lesion/site. Unequivocal progression of non-measurable disease in the opinion of the treating physician (an explanation must be provided). Death due to disease without prior documentation of progression. PFS is measured from date of registration to date of first observation of progressive disease, or death due to any cause. Patients last known to be alive and progression-free are censored at date of last contact.
Time Frame: 0-2 years
Population: All eligible patients who started treatment were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R-CHOP + I-131-tositumomab
Number analyzed (Participants) | 84
percentage of participants | 69 [59 to 79]

2. Primary Outcome: Response Rate (Complete, Complete Unconfirmed, and Partial)
Description: Complete Response(CR) is a complete disappearance of all disease with the exception of nodes. No new lesions. previously enlarged organs must have regressed and not be palpable. Bone marrow(BM) must be negative if positive at baseline. Normalization of markers. CR Unconfirmed (CRU) does not qualify for CR above, due to a residual nodal mass or an indeterminate BM. Partial Response(PR) is a 50% decrease in the sum of products of greatest diameters (SPD) for up to 6 identified dominant lesions, including spleenic and hepatic nodules from baseline. No new lesions and no increase in the size of liver, spleen or other nodes.
Time Frame: 6 months
Population: All eligible patients who started treatment were included in the analysis
Measure: Number; unit: participants
Arm/Group | R-CHOP + I-131-tositumomab
Number analyzed (Participants) | 84
participants
  Partial Response | 21
  Confirmed Response | 41
  Unconfirmed Response | 10
  No Response | 12

3. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: 6 months (assessed at the end of each cycle of chemotherapy for 8 cycles (1 cycle= 21 days), at restaging, and at the end of each radiolabeled antibody treatment)
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | R-CHOP + I-131-tositumomab
Number analyzed (Participants) | 84
Participants
  Anorexia | 2
  Calcium, serum-low (hypocalcemia) | 1
  Cardiac troponin I (cTnI) | 1
  Cardiac-ischemia/infarction | 3
  Constipation | 1
  Cough | 1
  Dehydration | 1
  Dizziness | 1
  Dyspnea (shortness of breath) | 2
  Fatigue (asthenia, lethargy, malaise) | 12
  Febrile neutropenia | 14
  Gastrointestinal-Other (Specify: GI bleed) | 1
  Glucose, serum-high (hyperglycemia) | 5
  Hearing: pts w/o audiogram not enroll monitor prgm | 1
  Hemoglobin | 12
  Hemorrhage, GI - Rectum | 1
  Hemorrhage, GU - Urinary NOS | 1
  Hypotension | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 2
  Inf (clin/microbio) w/Gr 3-4 neuts - Skin | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - UTI | 2
  Inf (clin/microbio) w/Gr 3-4 neuts - Upper airway | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Blood | 2
  Inf w/normal ANC or Gr 1-2 neutrophils - Dental | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 2
  Inf w/normal ANC or Gr 1-2 neutrophils - UTI | 1
  Left ventricular systolic dysfunction | 1
  Leukocytes (total WBC) | 47
  Lymphopenia | 39
  Mood alteration - anxiety | 1
  Muscle weakness, not d/t neuropathy - body/general | 1
  Nausea | 1
  Neurology-Other (Specify: restless leg syndrom) | 1
  Neuropathy: motor | 1
  Neuropathy: sensory | 8
  Neutrophils/granulocytes (ANC/AGC) | 55
  Opportunistic inf associated w/gt=Gr 2 lymphopenia | 2
  Pain - Abdomen NOS | 2
  Pain - Back | 1
  Pain - Esophagus | 1
  Pain - Head/headache | 1
  Phosphate, serum-low (hypophosphatemia) | 1
  Platelets | 29
  Pneumonitis/pulmonary infiltrates | 1
  Potassium, serum-low (hypokalemia) | 2
  Renal failure | 1
  Restrictive cardiomyopathy | 1
  SVT and nodal arrhythmia - Atrial fibrillation | 1
  SVT and nodal arrhythmia - SVT tachycardia | 1
  Secondary Malignancy-poss rel to cancer Tx | 2
  Sodium, serum-low (hyponatremia) | 1
  Thrombosis/thrombus/embolism | 2
  Uric acid, serum-high (hyperuricemia) | 1
  Vision-blurred vision | 1

ADVERSE EVENTS:
Time Frame: 6 months (assessed at the end of each cycle of chemotherapy for 8 cycles (1 cycle= 21 days), at restaging, and at the end of each radiolabeled antibody treatment)
Arm/Group | R-CHOP + I-131-tositumomab
Serious Adverse Events (participants affected / at risk) | 8/84
Other Adverse Events (participants affected / at risk) | 84/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R-CHOP + I-131-tositumomab (N=84)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Cardiac-ischemia/infarction (Cardiac disorders) | 2
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 1
Hemorrhage, GI - Upper GI NOS (Gastrointestinal disorders) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 1
Platelets (Investigations) | 1
Secondary Malignancy-poss rel to cancer Tx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Renal failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | R-CHOP + I-131-tositumomab (N=84)
Febrile neutropenia (Blood and lymphatic system disorders) | 13
Hemoglobin (Blood and lymphatic system disorders) | 70
Vision-blurred vision (Eye disorders) | 5
Constipation (Gastrointestinal disorders) | 40
Diarrhea (Gastrointestinal disorders) | 22
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 7 — Fluid--filled hiatal hernia in chest, causes reflux, GI bleed, Stomach upset, sore throat, Indigestion
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 15
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 45
Pain - Abdomen NOS (Gastrointestinal disorders) | 20
Pain - Oral cavity (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 12
Constitutional Symptoms-Other (Specify) (General disorders) | 6 — Sore throat, running nose, feeling cold, expressed as "post traumatic stress", Feels :groggy" from the vicodin
Edema: head and neck (General disorders) | 5
Edema: limb (General disorders) | 20
Fatigue (asthenia, lethargy, malaise) (General disorders) | 72
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 18
Pain-Other (Specify) (General disorders) | 11 — Pain noted in L upper quadrant, Few episodes once initiated G-CSF in sternal area, Intermittent heel and bilateral plantar burning, Chest pain, Pain in foot and ankle, toenail pain, Jaw, Occasional phantom pain in left groin
Rigors/chills (General disorders) | 11
Allergic reaction/hypersensitivity (Immune system disorders) | 9
Inf w/normal ANC or Gr 1-2 neutrophils - Sinus (Infections and infestations) | 5
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 20
AST, SGOT (Investigations) | 27
Alkaline phosphatase (Investigations) | 13
Creatinine (Investigations) | 18
Leukocytes (total WBC) (Investigations) | 70
Lymphopenia (Investigations) | 54
Metabolic/Laboratory-Other (Specify) (Investigations) | 8 — elevated LDH, increased blood urea nitrogen
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 68
Platelets (Investigations) | 62
Weight gain (Investigations) | 6
Weight loss (Investigations) | 19
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 18
Anorexia (Metabolism and nutrition disorders) | 23
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 11
Dehydration (Metabolism and nutrition disorders) | 6
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 47
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 8
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 10
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 9
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 15
Pain - Back (Musculoskeletal and connective tissue disorders) | 15
Pain - Bone (Musculoskeletal and connective tissue disorders) | 18
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 5
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 13
Pain - Joint (Musculoskeletal and connective tissue disorders) | 14
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 12
Dizziness (Nervous system disorders) | 18
Neuropathy: motor (Nervous system disorders) | 5
Neuropathy: sensory (Nervous system disorders) | 48
Pain - Head/headache (Nervous system disorders) | 22
Taste alteration (dysgeusia) (Nervous system disorders) | 17
Insomnia (Psychiatric disorders) | 23
Mood alteration - agitation (Psychiatric disorders) | 5
Mood alteration - anxiety (Psychiatric disorders) | 18
Mood alteration - depression (Psychiatric disorders) | 13
Urinary frequency/urgency (Renal and urinary disorders) | 8
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 24
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 23
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary/Upper Respiratory-Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 7 — Bronchiectasis from childhood exacerbated by chemotherapy, mild sore throat and some upper respiratory symptoms, crackles, decreased breath sounds, tachypnea, nasal congection
Dermatology/Skin-Other (Specify) (Skin and subcutaneous tissue disorders) | 8 — Actinic keratosis, Some sun damage on face, heavily freckled, erythema on ears, side of face; reaction to Rituximab, Appears pale, excoriated skin lesion
Dry skin (Skin and subcutaneous tissue disorders) | 6
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 51
Nail changes (Skin and subcutaneous tissue disorders) | 6
Pruritus/itching (Skin and subcutaneous tissue disorders) | 5
Rash/desquamation (Skin and subcutaneous tissue disorders) | 13
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 5
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 14
Hypotension (Vascular disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No